CLINICAL TRIAL: NCT04715425
Title: Thoracoscopic Surgical Versus Catheter Ablation Approaches for Primary Treatment of Persistent Atrial Fibrillation
Acronym: APPROACH AF
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Academisch Medisch Centrum - Universiteit van Amsterdam (AMC-UvA) (Other)
Responsible Party: Principal Investigator, J.R. de Groot, prof. dr. J.R. de Groot, Academisch Medisch Centrum - Universiteit van Amsterdam (AMC-UvA)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NL63978.018.18
Record Dates: First submitted 2021-01-13; First posted 2021-01-20 (Actual); Last update posted 2024-01-25 (Actual); Status verified 2024-01

CONDITIONS: Atrial Fibrillation, Persistent
Keywords: Catheter ablation; Thoracoscopic ablation
MeSH Terms: conditions — Atrial Fibrillation | interventions — Amputation, Surgical

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Thoracoscopic ablation (Active Comparator): Thoracoscopic ablation
  Interventions: Procedure: Thoracoscopic pulmonary vein isolation without additional lesion + left atrial appendage exclusion/amputation
- Catheter ablation (Active Comparator): Catheter ablation
  Interventions: Procedure: Catheter pulmonary vein isolation without additional lesions

INTERVENTIONS:
Procedure: Thoracoscopic pulmonary vein isolation without additional lesion + left atrial appendage exclusion/amputation — Bilateral pulmonary vein isolation using radiofrequency energy
  Arms: Thoracoscopic ablation
Procedure: Catheter pulmonary vein isolation without additional lesions — Bilateral pulmonary vein isolation using radiofrequency energy
  Arms: Catheter ablation

SUMMARY:
Rationale: Atrial fibrillation (AF) is a highly prevalent cardiac arrhythmia. AF is classified as paroxysmal or persistent AF, based on the duration and persistency of the arrhythmia. Despite state-of-the-art pharmacological therapies targeting the ventricular rate or aiming to restore sinus rhythm, many patients with persistent AF stay symptomatic. Catheter ablation, endocardial pulmonary vein isolation (PVI) in particular, is the most commonly applied approach to treat drug refractory persistent AF, but particularly in this patient group results are modest. Alternatively, the PVs can be approached epicardially by thoracoscopic surgery to isolate the PVs. This approach is more efficacious, at the cost of a more invasive procedure and longer hospital stay. However, no studies have been conducted comparing catheter with thoracoscopic ablation in patients with persistent AF as a primary invasive procedure after failing treatment with anti-arrhythmic medication.

Objective: This current study aims to assess a patient specific therapy plan for patients with persistent AF by randomizing thoracoscopic versus catheter ablation for PVI without adjuvant substrate ablation in those patients.

Study design: This is a prospective, non-blinded randomized multicenter study. Subjects will be randomized (1:1) to one of the two study-arms (thoracoscopic surgical or catheter PVI). The follow-up will last 5 years, with heart rhythm monitoring at three and six months, one year and yearly in the following years. In case AF recurs during the first year, the subject will receive the treatment of the otherother arm, or according to patient choice or clinical routine.

Study population: Patients with an indication for invasive treatment of persistent AF.

Intervention: Thoracoscopic surgical or catheter PVI without additional lesions.

ELIGIBILITY:
Inclusion Criteria:

* Age is between 18 and 80 years
* Persistent AF as defined following the ESC 2016 Guidelines, evidenced by 1) ongoing AF on the ECG or 2) documentation of AF necessitating cardioversion.
* AF documented by ECG or Holter < 1 year ago.
* At least one class I or III anti-arrhythmic drug in standard dosage has failed or is not tolerated.
* Left atrial volume index ≤ 45 ml/m2
* Legally competent and willing to sign the informed consent.
* Willing and able to adhere to the follow-up visit protocol.
* Life expectancy of at least 2 years.

Exclusion Criteria:

* Prior intervention (catheter ablation or minimally-invasive thoracoscopic ablation) for AF.
* AF is secondary to electrolyte imbalance, thyroid disease or other reversible or non-cardiovascular causes.
* Documentation of CTI dependent atrial flutter
* Valvular AF
* Paroxysmal AF
* Long standing Persistent AF, defined as AF continuously present for longer than 1 year.
* Body mass index >35kg/m2
* NYHA class IV heart failure symptoms or left ventricular ejection fraction <35%.
* NYHA class III heart failure symptoms, unless caused or aggravated by AF.
* Myocardial infarction within the preceding 2 months.
* Active infection or sepsis (as evidenced by increased white blood cell count, elevated CRP level or fever >38,5 °C).
* Known and documented carotid stenosis > 80%
* Planned cardiac surgery for other purposes than AF.
* Pregnancy or child bearing potential without adequate anticonception.
* Requirement of anti-arrhythmic drugs for ventricular arrhythmias.
* Presence of intracardiac mass or thrombus (discovery of any thrombus or intracardiac mass after signing of the informed consent will result in withdrawal of the subject from the study)
* Co-morbid condition that possesses undue risk of general anesthesia or port access cardiac surgery (in the opinion of the operator).
* History of previous radiation therapy on the thorax
* Circumstances that prevent follow-up
* No vascular access for catheterization.
* History of previous thoracotomy.
* Factors precluding transseptal puncture for catheterization.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 170 (Estimated)
Dates: Start 2019-09-25 (Actual); Primary Completion 2024-09 (Estimated); Study Completion 2028-09 (Estimated)

PRIMARY OUTCOMES:
Freedom of AF, defined as absence of any atrial tachyarrhythmia | Up until 72 patients experienced AF recurrence
  The primary endpoint of the study is freedom of AF, defined as absence of any atrial tachyarrhythmia without the use of antiarrhythmic drugs once a total number of 72 patients with AF recurrences after a single procedure have been reached. This is an event based endpoint. Freedom of atrial tachyarrhythmia is defined as the absence of documentation of episodes of atrial tachyarrhythmia lasting more than 30 seconds on Holter recordings during follow-up and/or on ECGs recorded outside the scope of the study.

SECONDARY OUTCOMES:
One year freedom of AF | 1 year of follow-up
  Freedom of arrhythmia with or without AAD after a single procedure after one year
Freedom of AF after two procedures | 1 year of follow-up after the second procedure
  Freedom of arrhythmia after 12 months with or without AAD after both procedures
Long term freedom of AF | 5 years of follow-up
  Freedom of arrhythmia after 5 years
Cost-effectiveness | 1 year of follow-up
  calculation of cost-effectiveness of both procedures in isolation, and the combination of both procedures.
Quality of life after a thoracoscopic surgical procedure or a catheter ablation procedure. | Yearly until 5 years follow-up
  Quality of life score of all patients, in both groups. We use the general (EQ5D) and AF specific (AFEQT) quality of life outcome questionaires.

CONTACTS AND LOCATIONS:
Locations (3):
- Netherlands (3):
  - Amsterdam University Medical Center location AMC, Amsterdam
  - Maastricht UMC+, Maastricht
  - St. Antonius Ziekenhuis Nieuwegein, Nieuwegein

IPD SHARING:
Plan to Share IPD: No